CLINICAL TRIAL: NCT02518451
Title: Bioequivalence Study of 160 mg Valsartan Film-coated Caplets Produced by PT Dexa Medica in Comparison With the Innovator Film-coated Tablets (Diovan® 160, Novartis Pharma AG)
Brief Title: Bioequivalence Evaluation of Two Film-Coated Formulations of Valsartan 160 mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PR. 183/EQL/2010
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: antihypertensive; bioequivalence; formulation; pharmakokinetic; valsartan; subjects; Fasting conditions
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- (Test) Group I (Experimental): Valsartan 160 mg film-coated caplets of PT Dexa Medica
  Interventions: Drug: Valsartan 160 mg film-coated caplets (test formulation)
- (Reference) Group II (Active Comparator): Valsartan 160 mg film-coated caplets (Diovan® 160)
  Interventions: Drug: Valsartan 160 mg film-coated caplets (reference formulation)

INTERVENTIONS:
Drug: Valsartan 160 mg film-coated caplets (test formulation) — In each of the two study periods (separated by a washout of one week) a single dose of test or reference formulation was administered.
  Other Names: Valsartan 160 mg of PT Dexa Medica
  Arms: (Test) Group I
Drug: Valsartan 160 mg film-coated caplets (reference formulation) — In each of the two study periods (separated by a washout of one week) a single dose of test or reference formulation was administered.
  Other Names: Diovan® 160
  Arms: (Reference) Group II

SUMMARY:
This was a randomized, single-blind, two-period, two sequence cross-over study under fasting condition, with a one-week wash-out period, to compare the pharmacokinetic profiles and bioavailability of two formulations (the test and reference) of valsartan 160 mg film-coated caplets.

DETAILED DESCRIPTION:
In the first period, subjects received either the test formulation (160 mg valsartan film-coated caplets produced by PT Dexa Medica, Palembang, Indonesia) once daily, or the innovator film-coated tablets (Diovan® 160, Novartis Farmaceutica S.A., Barbera del Valles, Spain for Novartis Pharma AG, Basel, Switzerland) once daily as the reference formulation. In the subsequent period, after a one-week wash-out period, they received the alternate drug.

At the night before starting the study, subjects were instructed to fast from any food and drink but mineral water for 9 hours before the drug administration. In the morning after, at the dosing day, each of the 48 subjects then swallowed (without chewing) one dose of valsartan 160 mg of the test formulation or of the reference formulation, with 200 mL of water. As much as 5 mL of blood samples for drug assay were drawn again from each subject, at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 9, 12, 16, 24, 36, and 48 hours after dosing.

The concentrations of valsartan in plasma were assayed using a validated high performance liquid chromatography with fluorescence detector (HPLC-FL) method. Pharmacokinetic parameters, including the area under the concentration-versus-time curve (AUC) from time zero to the time of last quatifiable concentration (48 hours after dosing) (AUC-t), AUC from time zero extrapolated to infinity (AUC-inf), maximum concentration (Cmax), time to reach the maximum concentration (tmax), and half-life (t1/2), were assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening.
2. Aged 18 - 55 years inclusive
3. Preferably non-smokers or smoke less than 10 cigarettes per day.
4. Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study.
5. Body mass index within 18 to 25 kg/m2.
6. Vital signs (after 10 minutes rest) must be within the following ranges:

   * Systolic blood pressure : 110 - 120 mm Hg
   * Diastolic blood pressure : 70 - 80 mm Hg
   * Pulse rate : 60 - 90 bpm

Exclusion Criteria:

1. Personal/family history of allergy or hypersensitivity or contraindication to valsartan or allied drugs.
2. Pregnant or lactating women (urinary pregnancy test will be applied to women subjects just before taking the study drug).
3. Any major illness in the past 90 days or clinically significant ongoing chronic medical illness e.g. congestive heart failure, hepatitis, hypotensive episodes, hyperglycemia, etc.
4. Presence of any clinically significant abnormal values during screening e.g. significant abnormality of liver function test (ALT, alkaline phosphatase, total bilirubin >= 1.5 ULN), renal function test (serum creatinine concentration > 1.4 mg/dL), etc.
5. Positive Hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV.
6. Clinically significant haematology abnormalities.
7. Clinically significant electrocardiogram (ECG) abnormalities.
8. Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism or excretion of the study drug, e.g. gastrointestinal diseases including gastric or duodenal ulcers or history of gastric surgery.
9. Past history of anaphylaxis or angioedema.
10. History of drug or alcohol abuse within 12 months prior to screening for this study.
11. Participation in any clinical trial within the past 90 days calculated from the last visit.
12. History of any bleeding or coagulative disorders.
13. History of difficulty with donating blood or difficulty in accessibility of veins in left or right arm.
14. A donation or loss of 300 mL (or more) of blood within 3 months before this study's first dosing day.
15. Intake of any prescription or non-prescription drug, food supplement or herbal medicine within 14 days of this study's first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
AUCt | 48 hours
  Area under the curve of plasma concentrations versus time from time zero to the time of last observed quantifiable concentration was determined from plasma concentration of two valsartan160 mg film-coated caplets formulations (test and reference formulations)
AUCinf | 48 hours
  Area under the curve of plasma concentrations versus time from time zero to infinity was determined from plasma concentration of two valsartan160 mg film-coated caplets formulations (test and reference formulations)
Cmax | 48 hours
  The maximum (peak) plasma concentration was determined from plasma concentration of two valsartan160 mg film-coated caplets formulations (test and reference formulations)

SECONDARY OUTCOMES:
Tmax | 48 hours
  The time of peak plasma concentration was determined from plasma concentration of two valsartan160 mg film-coated caplets formulations (test and reference formulations)
T1/2 | 48 hours
  The elimination half-life was determined from plasma concentration of two valsartan160 mg film-coated caplets formulations (test and reference formulations)

OTHER OUTCOMES:
Adverse events | 1 months
  The presence of adverse events will be observed, reported and sufficiently handled during subjects' participation in the study (1 month).

CONTACTS AND LOCATIONS:
Overall Officials: Effi Setiawati, MSc, Study Director — PT Equilab International
Locations (1):
- PT Equilab International, Jakarta, Jakarta Special Capital Region, Indonesia